CLINICAL TRIAL: NCT02261480
Title: Investigation in Sickle Cell Disease of a New Reagent Assay Examining Natural Parvovirus B19 Infection
Brief Title: A New Reagent Assay Examining Natural Parvovirus B19 Infection in Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: iSCREEN
Record Dates: First submitted 2014-10-06; First posted 2014-10-10 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Sickle Cell Disease
Keywords: Parvovirus B19 Infection
MeSH Terms: conditions — Anemia, Sickle Cell; Erythema Infectiosum | interventions — Blood Specimen Collection; Nasal Lavage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and/or nasopharyngeal wash samples will be taken and retained. If participants agree, leftover samples will be saved for potential health research in the future.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group A: Documented Prior History: Pediatric and adult participants with sickle cell disease (SCD) with a documented prior history of parvovirus B19 infection (aplastic crisis).
  Group A participants will have blood draw and nasopharyngeal wash on day 1 only. Nasopharyngeal wash will be optional for Group A.
  Interventions: Other: Blood draw; Other: Nasopharyngeal wash
- Group B: No Prior History: Pediatric and adult participants with SCD who have never had a documented parvovirus B19 infection (aplastic crisis).
  Group B participants will have blood draw and nasopharyngeal wash on day 1 only. Nasopharyngeal wash will be optional for Group B.
  Interventions: Other: Blood draw; Other: Nasopharyngeal wash
- Group C: Suspected and/or Confirmed: Sickle cell disease patients with suspected and/or confirmed acute parvovirus B19 infection, the latter defined as febrile illness with anemia without adequate compensatory reticulocytosis.
  Group C participants will have blood draw and nasopharyngeal wash on day 1, day 7±4 days, day 30±7 days, and day 120±14 days.
  Interventions: Other: Blood draw; Other: Nasopharyngeal wash

INTERVENTIONS:
Other: Blood draw — When possible, blood will be drawn as an extra aliquot utilizing the same needle stick procedure performed for standard of care.
Other: Nasopharyngeal wash — Nasopharyngeal washes are optional for Group A and Group B participants. Nasopharyngeal washes will be performed on all subjects in Group C. The technique used will be the same as used for regular standard of care per St. Jude guidelines.

SUMMARY:
Parvovirus B19 is a small virus that is the cause of "fifth" disease, a common infection in childhood. In people with sickle cell disease (SCD), parvovirus B19 infection causes the bone marrow to stop producing red blood cells temporarily, which can be life-threatening. A novel vaccine is currently in development for children with SCD. This study is the first step within a larger parvovirus B19 multi-institutional project that will help develop this new vaccine, as it will define the value and utility of using a novel assay for measurement of parvovirus-specific antibodies. The main objective is to investigate the relationship between the newly developed VP1u ELISA assay and the gold standard neutralization assay for parvovirus B19 infection.

The most accurate test, called a neutralizing antibody assay, to see if a person has had or currently has the infection is very complex and expensive and would be very difficult to use in a large research study to test the new vaccine. A new and simpler test has developed. The main goal of this study, iSCREEN, is to find out if this new test works.

There will be distinct labs performing the VP1u ELISA and the neutralization assays and the respective laboratories will not have access to each other's results for individual subjects. The VP1u ELISA will be performed at St. Jude Children's Research Hospital. Neutralization assays will be conducted at the National Heart, Lung and Blood Institute.

DETAILED DESCRIPTION:
Participants with sickle cell disease (SCD) will be divided into three study groups depending on their history of parvovirus B19 infection. Each will have blood drawn and/or nasopharyngeal wash which will provide the biological material for evaluation by assay.

* Group A participants will have a documented prior history of parvovirus B19 infection (aplastic crisis).
* Group B participants will have no documented history of parvovirus B19 infection (aplastic crisis) and will serve as the negative controls for the investigation of the relationship between the VP1u ELISA and the gold standard neutralization assay for parvovirus B19 infection.
* Group C participants will have suspected and/or confirmed acute parvovirus B19 infection (febrile illness with anemia without adequate compensatory reticulocytosis).

PRIMARY OBJECTIVES

* To estimate the correlation between the VP1u enzyme-linked immunosorbent assay (ELISA) and the gold standard neutralization assay for parvovirus B19 infection in subjects with SCD who have had a documented infection from parvovirus B19 causing aplastic crisis.
* To identify a cut-off for negativity in the VP1u ELISA and in the neutralization assay in subjects with SCD.

SECONDARY OBJECTIVES

* To characterize the performance characteristics of the VP1u ELISA, including sensitivity and specificity.
* To describe the kinetics of antibody responses generated following an acute parvovirus B19 infection in the serum and in the nasal mucosa of patients with SCD.

ELIGIBILITY:
Inclusion Criteria - Individuals not experiencing an acute illness (Group A):

* Males and females with a diagnosis of SCD of any genotype
* Ages > 1 year.
* Medical records available for verification of prior parvovirus B19 infection status.

Exclusion Criteria - Individuals not experiencing an acute illness (Group A):

* Patients on chronic transfusion therapy.
* Patients experiencing an acute febrile illness.
* Any medical or social reason, which in the opinion of the principal investigators (PIs) would make the participation of the subject ill-advised.

Inclusion Criteria - Individuals with confirmed (Group B) or suspected (Group C) acute parvovirus B19 infection:

* Males and females with a diagnosis of SCD of any genotype.
* Ages > 1 year.
* Symptoms of acute parvovirus infection (defined as worsened anemia with insufficient compensatory reticulocytosis in the setting of a febrile illness).

Exclusion Criteria - Individuals with confirmed (Group B) or suspected (Group C) acute parvovirus B19 infection:

* Patients on chronic transfusion therapy.
* Current epistaxis
* Any medical or social reason, which in the opinion of the principal investigators (PIs) would make the participation of the subject ill-advised.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sickle cell disease patients being seen at St. Jude Children's Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Correlation between the new VP1u ELISA and neutralizing antibodies tests in participants with documented parvovirus B19 infection | Baseline
Mean assay value using new VP1u ELISA and neutralization assays between Group B and Group A participants | Baseline
  To identify the cut-off for negativity for this patient population in the VP1u ELISA and in the neutralization assays, an ROC analysis will be conducted.

SECONDARY OUTCOMES:
Compare the sensitivity and specificity of the VP1u ELISA with the neutralization assay | Baseline
  Sensitivity and specificity of VP1u ELISA will be assessed by using the neutralization assay as the gold standard.
Antibody response following acute parvovirus B19 infection | Baseline, and Days 7, 30 and 120
  Descriptive statistics, such as mean, standard deviation, median and range, will be developed and plotted.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Hankins, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols